CLINICAL TRIAL: NCT07337538
Title: Evaluation of Two Mini-implant Diameters in the Infra-zygomatic Crest Region (Split-mouth Randomized Clinical Trial)
Brief Title: Evaluation of Two Mini-implant Diameters in the Infra-zygomatic Crest Region.
Acronym: TADs
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Baghdad (Other)
Responsible Party: Principal Investigator, Ali Jabbar Al Ameri, student researcher, University of Baghdad
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Device Feasibility
Other Study IDs: 1152425
Record Dates: First submitted 2026-01-01; First posted 2026-01-13 (Actual); Last update posted 2026-01-20 (Actual); Status verified 2026-01

CONDITIONS: Implant Stability
Keywords: temporary anchorage device stability; Tads; mini implant; miniscrew
MeSH Terms: conditions — Tietz syndrome

STUDY DESIGN:
Intervention Model Description: 20 participants will be enrolled. Each participant will receive two interventions concurrently, with a 1.6-mm diameter mini-implant placed on one infra-zygomatic crest and a 2.0-mm diameter mini-implant placed on the contralateral side. The side allocation of implant diameter will be randomized in an alternating manner (left-right).
Who Masked: Participant
Masking Description: Participants will be blinded to the diameter of the mini-implants placed on each side. The investigator performing the insertion will not be blinded due to the obvious difference in implant diameter.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- 1.6 mm (Experimental): 1.6 x12 mm mini implant inserted in the infrazygomatic crest region according to split mouth allocation.
  Interventions: Device: insersion of two diameters of mini implant.
- 2 mm (Experimental): 2 x12 mm mini implant inserted in the infrazygomatic crest region according to split mouth allocation.
  Interventions: Device: insersion of two diameters of mini implant.

INTERVENTIONS:
Device: insersion of two diameters of mini implant. — insertion of the two diameters in the infrazygomatic crest region (IZC) bilaterally (one for each side) then check difference in primary stability, secondary stability, pain perception and failure rate.

SUMMARY:
The goal of this clinical trials is to compare two diameters, 1.6 and 2 mm, of mini implants both are 12 mm length placed in the infrazygomatic crest region. The main questions it aims to answer are:

which diameter is more suitable for IZC region 1.6 or 2mm in terms of primary stability, secondary stability, pain perception and failure rate.

20 participant will receive 40 mini implant bilaterally (20 in one side of 1.6mm, the other side 20 of 2mm).

participants will be asked to record visual analog scale (VAS) for 3 nights monitored monthly by the investigator.

DETAILED DESCRIPTION:
Using 1.6x12mm and 2x12mm of mini implants in the IZC area and measuring primary stability, secondary stability, failure rate and pain perception.

The primary stability will be measured immediately after insertion using Easycheck device (Dentium, South Korea).

The secondary stability will be measured two months after insertion using the same device.

Failure is considered when the mini implant become loose, peri-implant inflammation or fallen after insertion, it will be checked monthly for six months.

pain perception will be recorded by patients using visual analog scale (VAS) score sheet 24 , 48, 72 hour after insertion.

Null hypothesis There is no significant difference between 1.6 and 2mm IZC mini implant diameters in terms of primary stability, secondary stability, failure rate and pain perception.

ELIGIBILITY:
Inclusion Criteria:

1. Individuals aged between 15 and 38 years.
2. Patients currently undergoing orthodontic treatment with fixed appliances who require mini-implant placement in the upper buccal posterior region (IZC) for full-arch distalization or en-masse retraction.
3. Patients willing and able to adhere to the study protocol.
4. Recommended for the use of bilateral mini-implants.

Exclusion Criteria:

* Syndromic conditions, facial trauma, or previous bone-related surgery.

Ages: 15 Years to 38 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 20 (Estimated)
Dates: Start 2026-01-14 (Actual); Primary Completion 2026-09-01 (Estimated); Study Completion 2026-11-01 (Estimated)

PRIMARY OUTCOMES:
primary stability | immediately after insertion
  primary stability measurement using easy check device (Dentium, south Korea) giving range of (1 - 100).
secondary stability | two month after insertion.
  secondary stability measurement using easy check device (Dentium, south Korea) giving range of (1 - 100).

SECONDARY OUTCOMES:
pain perception | after insertion 24 hour, 48 hour, 72 hour.
  using Visual Analogue Score (VAS) [1-10] higher score means higher pain.
Failure rate | monthly for six months after insertion.
  Failure is considered when the mini implant become loose, peri-implant inflammation or fallen after insertion.

CONTACTS AND LOCATIONS:
Overall Officials: Ali J. Al Ameri, BDS., Principal Investigator — University of Baghdad
Locations (2):
- Iraq (2):
  - Saydiya dental clinic, Baghdad, Baghdad Governorate
  - Baghdad university, Baghdad, Baghdad Governorate

IPD SHARING:
Plan to Share IPD: No